CLINICAL TRIAL: NCT00005005
Title: Clinical Trial of Parathyroid Hormone (PTH) and Alendronate in Combination in the Treatment of Osteoporosis
Brief Title: PaTH Study: Parathyroid Hormone and Alendronate for Osteoporosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dennis Black (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor-Investigator, Dennis Black, Prinicipal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N01 AR92245; N01AR002245-000 (NIH); NIAMS-045
Record Dates: First submitted 2000-03-24; First posted 2000-03-27 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Osteoporosis
Keywords: PTH; Alendronate; Parathyroid hormone; Osteoporosis; Postmenopausal
MeSH Terms: conditions — Osteoporosis | interventions — Alendronate

ARMS (4):
- 1 (Experimental): Participants will receive PTH for 1 year followed by alendronate for 1 year.
  Interventions: Drug: PTH; Drug: Alendronate
- 2 (Experimental): Participants will receive PTH and alendronate for 1 year followed by alendronate for 1 year.
  Interventions: Drug: PTH; Drug: Alendronate
- 3 (Experimental): Participants will receive alendronate for 2 years.
  Interventions: Drug: Alendronate
- 4 (Active Comparator): Participants will receive PTH for 1 year followed by placebo for 1 year.
  Interventions: Drug: PTH

INTERVENTIONS:
Drug: PTH
  Arms: 1; 2; 4
Drug: Alendronate
  Arms: 1; 2; 3

SUMMARY:
This 2-year study will test the effectiveness of combining parathyroid hormone (PTH) and alendronate for treating osteoporosis in postmenopausal women. Alendronate is a drug used to treat osteoporosis and primarily prevents bone loss, whereas PTH increases bone formation. We will treat the study participants either with PTH and alendronate, alendronate alone, or PTH alone. We will determine the effects of these treatments by looking for changes in bone mineral density in the hip and spine.

DETAILED DESCRIPTION:
The PaTH study is a 2-year, multicenter, double-blind, placebo-controlled trial to test the efficacy of combining hPTH (1-84) and alendronate for treating osteoporosis in postmenopausal women.

238 women were randomized between 55 and 85 years of age to receive either: (1) PTH for 1 year followed by alendronate for 1 year; (2) PTH and alendronate for 1 year followed by alendronate for 1 year; (3) alendronate for 2 years; or (4) PTH for 1 year followed by placebo for 1 year. The primary endpoints are changes in bone mineral density at several sites and changes in biochemical markers.

In addition, we will assess specific biochemical markers of bone turnover (e.g., osteocalcin, deoxypridinoline, N-telopeptide, bone-specific alkaline phosphatase and bone sialoprotein) to determine if they can predict the skeletal response to combination therapy. We will also determine whether PTH positively affects ultrasound measurements in the calcaneus.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 55 and 85 years
* Postmenopausal (have not had any menses in the last 5 years)
* Have a bone mineral density scan (DXA) that can be evaluated at the spine AND at the hip with a T-score equal to or below -2.5 at the spine or the femoral neck or total hip OR T-score equal to or below -2.0 at the spine or the femoral neck or total hip and have at least one of the following risk factors for fracture: (a) age > 65 years; (b) history of postmenopausal fracture (nonvertebral or vertebral); or (c) maternal history of hip fracture
* Willing and able to self-administer daily injections

Exclusion Criteria:

* Have used estrogen (oral or patch) for more than 1 month in the last 6 months or more than 12 months in the last 2 years
* History of more than 12 months of bisphosphonate use ever, or any use (> 4 weeks) within the past 12 months
* History of rhPTH (recombinant human PTH) use
* Any major life-threatening illnesses
* Type 1 or uncontrolled type 2 diabetes mellitus (defined as hemoglobin A1C > 10.0), or currently using insulin
* Vitamin D level < 15 nanograms/ml
* History of kidney disease (creatinine > 2.0 mg/dl)
* Renal insufficiency (creatinine clearance < 40 mg/min)
* Any history of kidney stones
* Any history of hypercalciuria or currently have urine calcium/creatinine >300 mg
* History of hypercalcemia, sarcoidosis, or hyperparathyroidism
* History of active or treated tuberculosis or other granulomatous disorders
* History of breast cancer, melanoma, or hematologic malignancy that has required treatment within the last 10 years
* History of bone cancer or any other metabolic bone disease that has required treatment within the last 10 years
* History of any other nonskin cancer that has required treatment within the last 10 years
* History of symptomatic esophageal reflux, achalasia or esophageal stricture
* Currently taking > 7.5 mg systemic prednisone or equivalent per day
* Currently using > two puffs, four times/day of inhaled steroids
* Currently taking anticoagulants or anticonvulsants
* Have used Calcitonin within the past 3 months
* Have used Raloxifene in the last 6 months or for more than 12 months in the last 2 years
* Have used Tamoxifen in the last 6 months or for more than 12 months in the last 2 years
* Have used fluoride for at least a month within the past 5 years
* Currently taking > 1000 IU/day vitamin D or vitamin D analogues or metabolites
* Currently taking thyroid hormone replacement AND have a TSH < 0.1mIU/L

Ages: 55 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 1999-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Changes in bone mineral density at several sites and changes in biochemical markers | Year 2

SECONDARY OUTCOMES:
Predictive value of specific biochemical markers of bone turnover | Year 2

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Black, PhD, Principal Investigator — University of California, San Francisco
Locations (4):
- United States (4):
  - Maine Center for Osteoporosis, Bangor, Maine
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Black DM, Greenspan SL, Ensrud KE, Palermo L, McGowan JA, Lang TF, Garnero P, Bouxsein ML, Bilezikian JP, Rosen CJ; PaTH Study Investigators. The effects of parathyroid hormone and alendronate alone or in combination in postmenopausal osteoporosis. N Engl J Med. 2003 Sep 25;349(13):1207-15. doi: 10.1056/NEJMoa031975. Epub 2003 Sep 20. PMID 14500804
- [Result] Black DM, Bilezikian JP, Ensrud KE, Greenspan SL, Palermo L, Hue T, Lang TF, McGowan JA, Rosen CJ; PaTH Study Investigators. One year of alendronate after one year of parathyroid hormone (1-84) for osteoporosis. N Engl J Med. 2005 Aug 11;353(6):555-65. doi: 10.1056/NEJMoa050336. PMID 16093464
- [Result] Bauer DC, Garnero P, Bilezikian JP, Greenspan SL, Ensrud KE, Rosen CJ, Palermo L, Black DM. Short-term changes in bone turnover markers and bone mineral density response to parathyroid hormone in postmenopausal women with osteoporosis. J Clin Endocrinol Metab. 2006 Apr;91(4):1370-5. doi: 10.1210/jc.2005-1712. Epub 2006 Jan 31. PMID 16449339
- [Result] Sellmeyer DE, Black DM, Palermo L, Greenspan S, Ensrud K, Bilezikian J, Rosen CJ. Hetereogeneity in skeletal response to full-length parathyroid hormone in the treatment of osteoporosis. Osteoporos Int. 2007 Jul;18(7):973-9. doi: 10.1007/s00198-007-0336-x. Epub 2007 Feb 28. PMID 17333451
- [Result] Antoniucci DM, Sellmeyer DE, Bilezikian JP, Palermo L, Ensrud KE, Greenspan SL, Black DM. Elevations in serum and urinary calcium with parathyroid hormone (1-84) with and without alendronate for osteoporosis. J Clin Endocrinol Metab. 2007 Mar;92(3):942-7. doi: 10.1210/jc.2006-1788. Epub 2006 Dec 12. PMID 17164314